CLINICAL TRIAL: NCT07107750
Title: Phase I Trial of Emavusertib (CA-4948) in Combination With Cisplatin, Gemcitabine, and Durvalumab in Patients With Untreated Advanced or Metastatic Biliary Tract Cancer
Brief Title: Emavusertib (CA-4948) in Combination With Cisplatin, Gemcitabine, and Durvalumab in Patients With Untreated Advanced or Metastatic Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202512063
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Biliary Tract Cancer; Metastatic Biliary Tract Carcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — CA-4948; Gemcitabine; Cisplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation Dose Level 0 (starting dose): Emavusertib + Gemcitabine + Cisplatin + Durvalumab (Experimental): * Treatment will be administered on a 21-day cycle.
  * Emavusertib will be self-administered at the assigned dose by mouth twice per day at approximately 12-hour intervals.
  * Cisplatin and gemcitabine will be administered intravenously on Days 1 and 8 for up to 8 total cycles as per standard of care. Up to 2 cycles of gemcitabine and cisplatin, with or without durvalumab, may be given off protocol prior to enrollment; therefore some patients may receive only 6 or 7 cycles of gemcitabine, cisplatin, and durvalumab in combination with emavusertib on study. Durvalumab will be administered IV on Day 1 of each cycle. Durvalumab will continue in combination with emavusertib as maintenance therapy starting with Cycle 9 (or earlier, if patient discontinues cisplatin and gemcitabine prior to Cycle 9).
  Interventions: Drug: Emavusertib; Drug: Gemcitabine; Drug: Cisplatin; Biological: Durvalumab
- Dose Escalation Dose Level -1: Emavusertib + Gemcitabine + Cisplatin + Durvalumab (Experimental): * Treatment will be administered on a 21-day cycle.
  * Emavusertib will be self-administered at the assigned dose by mouth twice per day at approximately 12-hour intervals.
  * Cisplatin and gemcitabine will be administered intravenously on Days 1 and 8 for up to 8 total cycles as per standard of care. Up to 2 cycles of gemcitabine and cisplatin, with or without durvalumab, may be given off protocol prior to enrollment; therefore some patients may receive only 6 or 7 cycles of gemcitabine, cisplatin, and durvalumab in combination with emavusertib on study. Durvalumab will be administered IV on Day 1 of each cycle. Durvalumab will continue in combination with emavusertib as maintenance therapy starting with Cycle 9 (or earlier, if patient discontinues cisplatin and gemcitabine prior to Cycle 9).
  Interventions: Drug: Emavusertib; Drug: Gemcitabine; Drug: Cisplatin; Biological: Durvalumab
- Dose Expansion: Emavusertib + Gemcitabine + Cisplatin + Durvalumab (Experimental): * Treatment will be administered on a 21-day cycle.
  * Emavusertib will be self-administered at the assigned dose by mouth twice per day at approximately 12-hour intervals.
  * Cisplatin and gemcitabine will be administered intravenously on Days 1 and 8 for up to 8 total cycles as per standard of care. Up to 2 cycles of gemcitabine and cisplatin, with or without durvalumab, may be given off protocol prior to enrollment; therefore some patients may receive only 6 or 7 cycles of gemcitabine, cisplatin, and durvalumab in combination with emavusertib on study. Durvalumab will be administered IV on Day 1 of each cycle. Durvalumab will continue in combination with emavusertib as maintenance therapy starting with Cycle 9 (or earlier, if patient discontinues cisplatin and gemcitabine prior to Cycle 9).
  Interventions: Drug: Emavusertib; Drug: Gemcitabine; Drug: Cisplatin; Biological: Durvalumab

INTERVENTIONS:
Drug: Emavusertib — Provided by Curis.
  Other Names: CA-4948
Drug: Gemcitabine — Standard of care.
  Other Names: Gemzar
Drug: Cisplatin — Standard of care.
  Other Names: Platinol
Biological: Durvalumab — Standard of care.
  Other Names: Imfinzi

SUMMARY:
Based on preclinical data from the Lim lab (WUSM), the investigators hypothesize that IRAK4 inhibition cripples tumor-intrinsic survival signaling and effectively overcomes the desmoplastic and immune-suppressive tumor microenvironment (TME) to render chemo- and immunotherapies effective in GI malignancy. Therefore, this trial is designed to evaluate the combination of emavusertib (CA-4948) and standard chemoimmunotherapy in untreated advanced or metastatic biliary tract cancer (BTC).

DETAILED DESCRIPTION:
The first part of the study will be dose escalation of emavusertib in combination with standard of care (SOC) cisplatin, gemcitabine, and durvalumab. Once the expansion dose of emavusertib is determined, the expansion part of the study will open. All patients will be treated with emavusertib in combination with SOC cisplatin, gemcitabine, and durvalumab for up to 8 total cycles. Patients may receive no more than 8 total cycles of gemcitabine and cisplatin for BTC. Up to 2 cycles of gemcitabine and cisplatin, with or without durvalumab, may be given off protocol prior to enrollment; therefore, some patients may only receive 6 or 7 cycles of gemcitabine, cisplatin, and durvalumab in combination with emavusertib on study. After 8 cycles, patients will discontinue cisplatin and gemcitabine and continue maintenance emavusertib and durvalumab.

ELIGIBILITY:
Inclusion Criteria:

* Advanced unresectable or metastatic histologically or cytologically confirmed adenocarcinoma of the biliary tract, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder carcinoma. Patients whose tumor have mixed histology but predominantly (>50%) adenocarcinoma are allowed.
* Measurable defined by RECIST v1.1.
* No prior systemic treatment for advanced unresectable or metastatic BTC with the following exceptions:

  * Neoadjuvant or adjuvant systemic therapy completed > 6 months from planned C1D1.
  * Up to two prior cycles of gemcitabine/cisplatin/anti-PD1 with no evidence of disease progression is allowed
* At least 18 years of age.
* ECOG performance status 0, 1, or 2
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN or ≤ 3 x IULN in patients with documented Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 2 x IULN, unless there are liver metastases in which case AST and ALT ≤ 5.0 x IULN
  * Creatinine clearance ≥ 35 mL/min by Cockcroft-Gault
  * INR ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤1.5 x IULN
* Creatinine phosphokinase (CPK) elevation at screening < Grade 2 (CPK < 2.5 x IULN).
* Patients on a cholesterol lowering statin must be on a stable dose with no dose changes within 3 weeks prior to study start.
* The effects of emavusertib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 90 days after completion of the study.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Current use or anticipated need for alternative, holistic, naturopathic, or botanical formulations used for the purpose of cancer treatment. Use of medical marijuana is permitted.
* A history of other malignancy with the exception of 1) malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease; 2) or known indolent malignancies that do not require treatment and will likely not alter the course of treatment of BTC in the opinion of the investigator
* History of allogeneic organ or stem cell transplant.
* Currently receiving any other investigational therapeutic agents. Investigational tracers related to imaging studies are allowed with a 7 day-washout.
* Clinically active CNS metastasis; treated and asymptomatic metastasis allowed at the discretion of the sponsor/investigator or site PI. Radiotherapy to the brain must be completed > 10 days prior to planned C1D1.
* Chemoradiation with curative intent within 6 months prior to C1D1 of study therapy.
* Palliative radiation therapy within 10 days prior to C1D1 of study therapy.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to emavusertib, gemcitabine, cisplatin, durvalumab, or other agents used in the study.
* Concomitant use of drugs with a known risk of causing prolonged QTc (with exception of Zofran if needed for supportive care) and/or Torsades de Pointes or a history of risk factors for Torsades de Pointes.
* Presence of interstitial lung disease or pneumonitis ≥ G2 at time of screening.
* Administration of a live attenuated vaccine within 30 days prior to C1D1
* QTc (Fridericia) >470ms on screening EKG.
* Gastrointestinal condition which could impair absorption of emavusertib or inability to ingest emavusertib in the opinion of the investigator.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia in the opinion of the investigator.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of C1D1.
* Patients with known HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines and in line with contraindicated concomitant medications is recommended.
* Participants with active, known, or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll after discussion with the sponsor-investigator or site PI.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study treatment except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease. Note: treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study treatment is permitted. Inhaled intranasal, intra-articular, and topical steroid uses are permitted.
* History of grade 3 or greater rhabdomyolysis that did not completely resolve.
* Patients are unwilling to adhere to the lifestyle guidance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2030-05-31 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of emavusertib in combination with gemcitabine, cisplatin, and durvalumab in patients with BTC as measured by incidences and types of adverse events | From consent through 30 days after last dose of study treatment (estimated to be 15 months)
  Graded using CTCAE version 5.0.
Dose escalation only: To determine an expansion dose for emavusertib in combination with gemcitabine, cisplatin, and durvalumab in patients with BTC. | Completion of cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
Progression-free rate (PFR) | At 6 months from start of treatment
  * Defined as the proportion of evaluable patients who are free of disease progression/recurrence at 6 months from the start of treatment.
  * Response and progression will be evaluated in this study using the revised international criteria (RECIST version 1.1) proposed by the RECIST committee as well as the modified iRECIST guidelines. Until radiographic progression based on RECIST 1.1, there is no distinct iRECIST assessment.
Disease control rate (DCR) | At 6 months from start of treatment
  * DCR is the proportion of patients with either complete response (CR), partial response (PR), or stable disease (SD) (with a duration of SD for 6 months).
  * Complete Response (CR): Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Overall response rate (ORR) | Through completion of treatment (estimated to be 14 months)
  * ORR = number of patients with complete response or partial response
  * Complete Response (CR): Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 38 months)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. The alive patients without progression are censored at the last follow-up.
  * Response and progression will be evaluated in this study using the revised international criteria (RECIST version 1.1) proposed by the RECIST committee as well as the modified iRECIST guidelines. Until radiographic progression based on RECIST 1.1, there is no distinct iRECIST assessment.
Overall survival (OS) | Through completion of follow-up (estimated to be 38 months)
  OS is defined as the duration of time from start of treatment to time of death from any cause. The alive patients are censored at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Aranha, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu